CLINICAL TRIAL: NCT00003831
Title: Randomized Trial of Mediastinal Lymph Node Sampling Versus Complete Lymphadenectomy During Pulmonary Resection in the Patient With N0 and N1 (Less Than Hilar) Non-Small Cell Carcinoma
Brief Title: Lymph Node Removal in Treating Patients With Stage I or Stage II Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z0030; CDR0000066988 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lymph node sampling (Experimental): Patients undergo pulmonary resection. No additional lymph nodes are removed. Patients are followed at 4, 6, 8, 12, 18, 24, and 36 months and then annually thereafter until death.
  Interventions: Procedure: conventional surgery
- Lymph node dissection (Active Comparator): Patients undergo removal of nearly all of the lymph nodes from the central part of the chest between the lungs, followed by pulmonary resection. Patients are followed at 4, 6, 8, 12, 18, 24, and 36 months and then annually thereafter until death.
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Procedure: conventional surgery

SUMMARY:
RATIONALE: Surgical removal of all lymph nodes in the chest may kill cancer cells that have spread from tumors in the lung. It is not yet known whether complete removal of all lymph nodes in the chest is more effective than removal of selected lymph nodes in treating patients who have stage I or stage II non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of complete removal of all lymph nodes in the chest with that of selected removal of lymph nodes during lung cancer surgery in treating patients who have stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare whether a complete mediastinal lymph node dissection versus mediastinal lymph node sampling improves overall survival of patients with N0 or non-hilar N1 non-small cell lung cancer undergoing resection.
* Compare these two methods with reference to identification of occult mediastinal lymph node involvement.
* Compare the effect of these two methods on operative time and duration of postoperative complications, including chest tube drainage and length of hospitalization for these patients.
* Compare the effect of these two methods on local recurrence free survival and local regional recurrence free survival of these patients.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study only if ALL of the following criteria apply:

Pre-operative:

1. Patient must be ≥18 years of age.
2. Patient must have an ECOG/Zubrod performance status of ≤ 3.
3. Patient must have tissue diagnosis of a clinically resectable T1 or T2, N0 or non-hilar N1, M0 NSCLC (squamous cell carcinoma, large cell carcinoma or adenocarcinoma including bronchoalveolar carcinoma) established prior to randomization. NOTE: A patient without a pre-operative tissue diagnosis, but with clinically suspected NSCLC that fits the above criteria is eligible provided the tissue diagnosis is confirmed intraoperatively.
4. Patient must have pre-operative imaging procedure, CT scan of the chest and upper abdomen to include liver and adrenal glands to determine eligibility, within 60 days of the date of the pulmonary resection.
5. Patient that has not had a mediastinoscopy should have no mediastinal adenopathy on the CT of the chest defined as no lymph node > 1 cm in the shortest axis.
6. Patient is a candidate for a complete resection of the carcinoma via pneumonectomy,lobectomy, bilobectomy, or anatomic segmentectomy with or without sleeve resection,as noted in the surgical plan.
7. Patient, or patient's legally acceptable representative, must provide a signed and dated Z0030-specific written informed consent prior to registration and any study-related procedures.
8. If patient is a survivor of a prior cancer, the following criteria are met:

   1. Patient has undergone potentially curative therapy for all prior malignancies,
   2. No evidence of any prior malignancies for at least 5 years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone),
   3. Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.

Intra-operative:

1. Patient with right-sided lesions must have at least nodal stations #2R, 4R, 7 and 10 R examined. If the nodes are found, they must be sampled and proven negative by frozen section.
2. Patient with left-sided lesions must have at least nodal stations #5, 6, 7 and 10L examined. If the nodes are found, they must be sampled and proven negative by frozen section.
3. Any other suspicious mediastinal or hilar nodes must be sampled and proven negative by frozen section. Levels 2, 4 and 7 need not be re-sampled if they were sampled at a mediastinoscopy done within 60 days of thehoracotomy.

Exclusion Criteria:

A patient will NOT be eligible for inclusion in this study if ANY of the following criteria apply:

1. Patient has N2 disease determined at pre-operative mediastinoscopy or on sampling.
2. Patient has T3 or T4 tumor.
3. Patient is having only a wedge resection performed for treatment.
4. Patient has received prior chemotherapy or radiotherapy for this cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1023 (Actual)
Dates: Start 1999-07; Primary Completion 2006-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years

SECONDARY OUTCOMES:
Disease-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Allen, MD, Study Chair — Mayo Clinic
Locations (74):
- United States (70):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Veterans Affairs Medical Center - Gainesville, Gainesville, Florida
  - Shands Cancer Center at the University of Florida, Gainesville, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Medical Center of Southwest Louisiana, Lafayette, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Rhode Island Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - St. Luke's Hospital, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - Creighton University School of Medicine, Omaha, Nebraska
  - Englewood Hospital Oncology Program, Englewood, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Louis Busch Hager Cancer Center at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Trinity Hospital, Minot, North Dakota
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Tri-Health Good Samaritan Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon
  - Westmoreland Regional Hospital, Greensburg, Pennsylvania
  - Jameson Memorial Hospital, New Castle, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburg Medical Center - Shadyside Hospital, Pittsburgh, Pennsylvania
  - Presbyterian-University Hospital, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - St. Clair Memorial Hospital, Pittsburgh, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Saint Thomas Hospital, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Australia (2):
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
- Canada (2):
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. A genomic strategy to refine prognosis in early-stage non-small-cell lung cancer. N Engl J Med. 2006 Aug 10;355(6):570-80. doi: 10.1056/NEJMoa060467. PMID 16899777 (Retraction: PMID 21366430 Potti A, Mukherjee S, Petersen R, Dressman HK, Bild A, Koontz J, Kratzke R, Watson MA, Kelley M, Ginsburg GS, West M, Harpole DH Jr, Nevins JR. N Engl J Med. 2011 Mar 24;364(12):1176)
- [Result] Fibla JJ, Cassivi SD, Brunelli A, Decker PA, Allen MS, Darling GE, Landreneau RJ, Putnam JB. Re-evaluation of the prognostic value of visceral pleura invasion in Stage IB non-small cell lung cancer using the prospective multicenter ACOSOG Z0030 trial data set. Lung Cancer. 2012 Dec;78(3):259-62. doi: 10.1016/j.lungcan.2012.09.010. Epub 2012 Oct 3. PMID 23040416
- [Result] Darling GE, Allen MS, Decker PA, Ballman K, Malthaner RA, Inculet RI, Jones DR, McKenna RJ, Landreneau RJ, Putnam JB Jr. Number of lymph nodes harvested from a mediastinal lymphadenectomy: results of the randomized, prospective American College of Surgeons Oncology Group Z0030 trial. Chest. 2011 May;139(5):1124-1129. doi: 10.1378/chest.10-0859. Epub 2010 Sep 9. PMID 20829340
- [Result] Darling GE, Allen MS, Decker PA, Ballman K, Malthaner RA, Inculet RI, Jones DR, McKenna RJ, Landreneau RJ, Rusch VW, Putnam JB Jr. Randomized trial of mediastinal lymph node sampling versus complete lymphadenectomy during pulmonary resection in the patient with N0 or N1 (less than hilar) non-small cell carcinoma: results of the American College of Surgery Oncology Group Z0030 Trial. J Thorac Cardiovasc Surg. 2011 Mar;141(3):662-70. doi: 10.1016/j.jtcvs.2010.11.008. PMID 21335122
- [Result] Allen MS, Darling GE, Pechet TT, Mitchell JD, Herndon JE 2nd, Landreneau RJ, Inculet RI, Jones DR, Meyers BF, Harpole DH, Putnam JB Jr, Rusch VW; ACOSOG Z0030 Study Group. Morbidity and mortality of major pulmonary resections in patients with early-stage lung cancer: initial results of the randomized, prospective ACOSOG Z0030 trial. Ann Thorac Surg. 2006 Mar;81(3):1013-9; discussion 1019-20. doi: 10.1016/j.athoracsur.2005.06.066. PMID 16488712